CLINICAL TRIAL: NCT05540717
Title: A Randomised, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of PQ Grass in Subjects With Seasonal Allergic Rhinitis and/or Rhinoconjunctivitis Induced by Grass Pollen Exposure
Brief Title: Efficacy and Safety of PQ Grass in Subjects With Seasonal Allergic Rhinitis and/or Rhinoconjunctivitis Induced by Grass Pollen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQGrass306; 2019-001517-16 (EudraCT Number)
Record Dates: First submitted 2022-09-01; First posted 2022-09-15 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Seasonal Allergic Rhinitis; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PQ Grass (Experimental): 6 subcutaneous injections of active treatment (900, 2700, 6000, 6000, 6000 and 6000 SU sequentially) to achieve a cumulative nominal dose of 27600 SU
  Interventions: Biological: PQ Grass
- Placebo (Placebo Comparator): 6 subcutaneous injections of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PQ Grass — Suspension for Injection
  Arms: PQ Grass
Biological: Placebo — Solution for injection
  Arms: Placebo

SUMMARY:
The PQGrass306 (G306) clinical trial is the pivotal Phase III efficacy clinical trial of PQ Grass.

The aim of the G306 pivotal clinical trial is to confirm the efficacy and safety of the optimal effective dose of PQ Grass 27600 SU. This will be determined through the measurements of the effect of PQ Grass on the symptoms of seasonal allergic rhinitis (SAR)/rhinoconjunctivitis and the use of relief medications to control these symptoms during the peak grass pollen season (GPS).

DETAILED DESCRIPTION:
Multi-centre, randomised, parallel group, double-blind, placebo-controlled clinical trial to confirm the efficacy and safety of the optimal effective dose of PQ Grass (27600 SU).

Randomized study subjects, in a randomisation ratio of 1:1, will receive either treatment with 6 injections of active treatment (900, 2700, 6000, 6000, 6000 and 6000 SU sequentially) to achieve a cumulative nominal dose of 27600 SU, or 6 injections of placebo prior to the onset of the grass pollen season (GPS).

The aim of the study is to confirm the efficacy and safety of the optimal effective dose of the PQ Grass 27600 SU dose. Efficacy will be determined through the measurements of the effect of PQ Grass on the symptoms of seasonal allergic rhinitis (SAR)/rhinoconjunctivitis and the use of relief medications to control these symptoms during the peak GPS.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the ICF (informed consent form) and in this clinical trial protocol and to attend required clinical trial visits.
2. Subject who has a signed and dated ICF.
3. Subject must be 18 to 65 years of age inclusive, at the time of signing the ICF.
4. Male or female.
5. Female subjects who are not of childbearing potential (defined as at least 12 months natural spontaneous amenorrhoea, or at least 6 weeks following surgical menopause/permanent sterilisation [hysterectomy, bilateral oophorectomy and bilateral salpingectomy]) or females of childbearing potential who agree to comply with the contraceptive requirements of the clinical trial protocol.
6. Good general health, as determined by the Investigator, based on a medical evaluation, including medical history, physical examination, mental status assessment and laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the clinical trial procedures.
7. Positive history of moderate to severe symptoms of SAR/rhinoconjunctivitis ascribed to grass (Pooideae) pollen exposure of at least 2 seasons duration, despite having received allergy pharmacotherapy (e.g., antihistamines, nasal corticosteroids, leukotriene modifiers, etc.) during the last 2 consecutive grass pollen seasons prior to the clinical trial, confirmed by subject records.

   Please note: Subjects with asthma may be included, but the asthma must be well controlled (according to current Global Initiative for Asthma [GINA] guidelines [GINA 2022]).
8. A positive SPT (skin prick test) to histamine (wheals [longest diameter] ≥3 mm) and a negative SPT to the negative control (wheal diameter = 0 mm) at screening.
9. A positive SPT for grass pollen (wheals [longest diameter] ≥3 mm).
10. Grass specific IgE (immunoglobulin E) class ≥2 as documented by an ImmunoCAP test at screening.
11. Forced expiratory volume in one second (FEV1) ≥70% of predicted, with a FEV1/forced vital capacity (FVC) ratio >75% and PEFR (peak expiratory flow rate) ≥70% of predicted at screening.

Exclusion Criteria:

1. Pregnant or lactating subject.
2. Presence of any medical history of moderate to severe allergy symptoms (verified by a positive SPT at screening or positive specific IgE [≥2] at screening) to any other seasonal allergen (other than grass) or perennial allergens.

   Exception: Period 1, Period 2 and Period 3 of the entire clinical trial will be conducted outside of the pollen season(s) of concern or perennial allergies are irrelevant due to avoidance measures (e.g., cats and dog allergy). Subjects with mild allergy symptoms (only) to any other allergen apart from grass may be included at the discretion of the Investigator. In countries in Europe where Bermuda grass is present, any medical history of moderate to severe allergy symptoms to Bermuda grass (verified by a positive SPT or positive specific IgE [Class ≥2]), will also represent a reason for exclusion as it will not be possible to conduct Period 1, Period 2 and Period 3 of the entire clinical trial outside of Bermuda grass pollen season. Albeit Bermuda grass being commonly defined as a grass, it belongs to the Poaceae family, while the sentence (other than grass) in Exclusion criterion #2 refers to grass of Pooideae subfamily (as defined in Inclusion criterion #7).
3. Subjects at US clinical trial sites in regions where southern grasses (Bahia grass, Bermuda grass or Johnson grass) are the dominant grasses and the main cause of grass allergy symptoms with a positive SPT to any of the 3 grasses (irrespective of the severity of symptoms).
4. Moderate to severe symptoms during the 3 years prior to Visit 1 to any other seasonal or perennial allergen not tested in the SPT done at screening that cannot be avoided during the Period 1 to Period 3 of the clinical trial and the symptoms of which may interfere with administration of treatment and/or impact the data collected.
5. Presence of any medical condition that may reduce the ability to survive a serious allergic reaction.
6. Presence of active systemic autoimmune disorder, systemic autoimmune disorders in remission or active organ specific autoimmune disorder.
7. Presence of active malignant neoplasia, severe cardiovascular disease (e.g., coronary artery disease, cardiac insufficiency, etc.), pulmonary insufficiency, severe psychiatric disorders or primary and secondary immunodeficiencies.
8. History of any other immunological disorder or other diseases (including, but not limited cardiovascular [including uncontrolled or inadequately controlled hypertension], gastro-intestinal, hepatic, renal, haematological, neurological, endocrine or pulmonary disease) that in the opinion of the Investigator may pose a safety risk or compromise the interpretation of efficacy of the clinical trial treatment.
9. Presence of severe or poorly controlled or uncontrolled asthma as defined by at least 1 of the following criteria:

   1. Severe asthma (as per the current GINA guidelines [GINA, 2022]).
   2. Uncontrolled or poorly controlled asthma as per the current GINA guidelines (GINA, 2022).
   3. Asthma that requires more than a daily dose above 800 μg of inhaled budesonide (or clinically comparable inhaled corticosteroid) as per the current GINA guidelines (GINA, 2022).
   4. History of 2 or more systemic corticosteroid courses within 6 months of screening or Visit 2 or 1 course of systemic corticosteroids within 3 months of screening or Visit 2 to treat asthma.
   5. Prior intubation/mechanical ventilation for asthma.
   6. Emergency room visit or hospitalisation for asthma in the 12 months prior to screening or Visit 2.
   7. Any history of a life-threatening asthma attack.
   8. FEV1 <70% of predicted or FEV1/FVC ≤75% or PEFR <70% of predicted with or without controller medications at screening or Visit 2.
10. Presence non-atopic rhinitis and/or rhino-sinusitis (with or without polyps).
11. Presence of nasal polyps and/or chronic sinusitis.
12. Presence of any acute or chronic ocular disorder, other than allergic conjunctivitis.
13. Eye surgery within the past 6 months.
14. Presence of any skin conditions (e.g., skin abnormalities, tattoos etc.), which might interfere with the interpretation of the SPT results.
15. Clinical history of Type I diabetes or poorly controlled Type II diabetes.
16. Moderate to severe upper or lower respiratory infections requiring medication within 14 days before screening (Visit 1) or Visit 2.
17. Presence of acute or chronic infection, fever or inflammation at screening or Visit 2.
18. Clinical history of severe systemic reaction or serious systemic reaction in response to AIT (allergen immunotherapy) in the past.
19. Clinical history of severe or life-threatening anaphylactic reactions to foods, insect venom, exercise, drugs or idiopathic anaphylaxis.
20. Clinical history of allergy, hypersensitivity or intolerance to the excipients of the investigational drug/placebo.
21. Clinical history of allergy, hypersensitivity or intolerance to the relief medications (for relief of allergy symptoms during Period 3) provided for use in this clinical trial.
22. Clinical history of hereditary angioedema.
23. Unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated such as in subjects with hyperthyroidism, uncontrolled hypertension, cardiac arrhythmias, closed angle glaucoma or subjects taking other sympathomimetics).
24. Tyrosine metabolism disorders, especially tyrosinemia and alkaptonuria.
25. Clinical history of drug or alcohol abuse, which, in the Investigator's opinion, could interfere with the subject's ability to participate in the clinical trial.
26. Subjects who have suspicion or symptoms of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (as assessed by the Investigator) or who have had unprotected contact with a confirmed case of COVID-19 (coronavirus disease 2019) in the 2 weeks prior to screening or Visit 2 (based on the Investigator's discretion).
27. Subjects who were hospitalised for COVID-19 within 6 months prior to screening or Visit 2.
28. Any history of AIT for grass pollen allergy in the past or history of AIT for any other type of allergy (excluding food allergy) in the past 5 years.
29. Inability to adhere to the washout periods listed in the protocol, with respect to screening and to refrain from using the medications indicated until after Visit 11.
30. Treatment with a preparation containing MPL (monophosphoryl lipid-A) (e.g., Cervarix, Shingrix, Fendrix) within 2 years prior to Visit 1 and until after completion of Visit 11 (with the exception of the investigational drug).
31. Previous history of epinephrine auto-injector use.
32. β-blocker medication (local or systemic, including eye drops) for any indication.
33. Monoamine oxidase inhibitors and tricyclic antidepressants. Please note: Tricyclic antidepressants should be avoided at least 2 weeks prior to screening.
34. Any previous therapy (within the previous 5 years) or current therapy with anti IgE (e.g., omalizumab [Xolair]) or anti-interleukins (e.g., mepolizumab).
35. Current or past therapy (within the previous 5 years) with any other immunomodulatory biologics.
36. Unable to refrain from any vaccination (including influenza vaccine and COVID-19 vaccine) during the clinical trial (unless administered >30 days prior to randomisation).

    Please note: Emergency vaccinations (e.g., tetanus due to injury) can be administered at any time. Booster vaccinations (only) for COVID-19 can be administered during the clinical trial apart from during the treatment period. There should be at least 14 days interval from the last administration of the investigational drug/placebo prior to administration of a COVID-19 booster injection.
37. Participation in a clinical research trial with any investigational drug within 4 weeks of Visit 1 or concomitantly with this clinical trial.

    Please note: The period of exclusion begins at the time of the last visit of the prior clinical research trial. Subjects consented and screened, but not dosed in the prior clinical research trial are not excluded.
38. Personal, financial or other dependent relationship (e.g., employee or immediate relative) with the clinical trial site, Sponsor, Sponsor's representative, or another individual who has access to the clinical trial protocol.
39. Vulnerable subjects or those in judicial or governmental detention, detainment or imprisonment in a public institution.
40. Subjects likely to have prolonged periods of absence (e.g., business or personal travel) during the GPS defined as:

    * Absence of a total of 22 days or more in similar geographical regions (as determined by the Investigator), with no single trip in a similar geographical region exceeding 14 days.
    * Absence of a total of 15 days or more in non-similar geographic regions (as determined by the Investigator), with no single trip in a non-similar geographical region exceeding 7 days.
41. Have changed residence to a different geographical region(s) since the last GPS.

Exception: The old and new residences are in the same or similar geographical region as determined by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (33):
  - IMMUNOe Research Centers, Centennial, Colorado
  - Velocity Clinical Research Denver, Denver, Colorado
  - Allergy Partners of Central Kentucky, Lexington, Kentucky
  - Allergy and Asthma Associates of Bluegrass, Lexington, Kentucky
  - Family Allergy Asthma Research Institute, Louisville, Kentucky
  - Allergy & Asthma Specialists PSC, Owensboro, Kentucky
  - Northern Light Allergy and Immunology, Bangor, Maine
  - Paul A. Shapero M.D., Bangor, Maine
  - Chesapeake Clinical Research Inc, White Marsh, Maryland
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research of The Ozarks Inc - Warrensburg, Columbia, Missouri
  - Montana Medical Research, Missoula, Montana
  - Nebraska Medical Research Institute, The Asthma & Allergy Center, Bellevue, Nebraska
  - Parikh Institute for Research LLC, Highland Park, New Jersey
  - Atlantic Research Center LLC, Ocean City, New Jersey
  - Weiss Medical, Riverdale, New Jersey
  - Allergy Asthma and Immunology Research Institute, Charlotte, North Carolina
  - Cincinnati Allergy and Asthma Center, Cincinnati, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Optimed Research Ltd, Columbus, Ohio
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, LLC - CRN - PPDS, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Inc, Grants Pass, Oregon
  - Velocity Clinical Research - Medford - ERN - PPDS, Medford, Oregon
  - Northwest Research Center, Portland, Oregon
  - Allergy & Asthma Specialists, Blue Bell, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Allergy Associate of Utah, Murray, Utah
  - Lysosomal Rare Disorders Research & Treatment Center, Fairfax, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Bellingham Asthma Allergy and Immunology Clinic, Bellingham, Washington
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Austria (4):
  - Medizinische Universitaet Innsbruck - Universitatsklinik fuer Dermatologie, Venerologie und Allergologie, Innsbruck
  - Bezirkskrankenhaus Kufstein, Kufstein
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
  - Ambulatorium für Allergie und klinische Immunologie AAKI, Vienna
- Czechia (9):
  - Fakultní nemocnice u sv. Anny v Brně, Brno
  - MUDr. Jana Poloniová - alergologie a klinická imunologie, České Budějovice
  - Alergopraktik, s.r.o., Jablonec nad Nisou
  - Alergologie a imunologie MUDr. Hofstetr, Jihlava
  - Alergoimuno s.r.o., Ostrava-Hrabuvka
  - ACREDULA BENEDICTA s.r.o., Pardubice
  - Fakultní nemocnice Plzeň, Pilsen
  - KASMED, s.r.o., Tábor
  - MŮJ ALERGOLOG s.r.o., Trutnov
- Germany (29):
  - CIMS Studienzentrum Bamberg, GmbH, Bamberg
  - Charité - Universitaetsmedizin Berlin Klinik fuer Dermatologie, Venerologie und Allergologie/ Abteilung Allergologie und Immunologie, Berlin
  - Praxis Dr. Petra El-Naib, Chemnitz
  - HNO-Praxis Dr. Udo Schaefer, Dresden
  - Klinische Forschung Dresden GmbH, Dresden
  - Praxis fuer HNO und Allergologie, Dresden
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - HNO-Praxis Dr. Uta Thieme, Duisburg
  - RKM740 Hals-Nasen-Ohrenheilkunde, Düsseldorf
  - Gemeinschaftspraxis Ruhr, Essen
  - Medizentrum Essen Borbeck, Essen
  - Medaimun GmbH, Frankfurt am Main
  - medicoKIT GmbH, Goch
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Hamburger Institut für Therapieforschung GmbH, Hamburg
  - Velocity Clinical Research Hamburg, Hamburg
  - Praxis Dres. med. Florian Heimlich und Angelika Witzel-Heimlich, Heidelberg
  - HNO-Praxis Landsberg, Landsberg
  - Praxis fuer Pneumologie und Allergologie, Leipzig
  - Sektion Rhinologie/Allergologie Klinik fuer HNO-Heilkunde, UKGM - Marburg, Marburg
  - Beldio Research GmbH, Memmingen
  - Facharztpraxis Dr. med. Jan-Christof Bohn, Mittweida
  - Ballenberger, Freytag, Wenisch Institut fuer klinische Forschung GmbH, Neu-Isenburg
  - Studienzentrum Maerkisch-Oderland, Neuenhagen
  - KliFOs - Klinische Forschung Osnabrueck, Osnabrück
  - Studienzentrum Dr. Sabine Lassmann, Saalfeld
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Klinikum Stuttgart - Krankenhaus Bad Cannstatt (KBC) - Frauenklinik, Stuttgart
  - Dres. med. Josef und Wilma Grosskopf, Wallerfing
- Hungary (4):
  - Gróf Tisza István Kórház Rendelőintézet MEDIDOCUMENT Kereskedelmi és Szolgáltató Betéti Társaság, Berettyóújfalu
  - Clinexpert Kft, Budapest
  - HiTech Medical Kft., Budapest
  - Pecsi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Pécs
- Poland (23):
  - Prywatny Gabinet Internistyczno - Alergologiczny, Bialystok
  - Allergy Clinic Homeo Medicus, Bialystok
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa
  - Centrum Medyczne Pratia Katowice, Katowice
  - Specjalistyczna Praktyka Lekarska dr n. med. Joanna Orlicz-Widawska, Katowice
  - ETG Kielce, Kielce
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o., Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Uniwersytecki Szpital Kliniczny im. Barlickiego, Poradnia alergologii i chorob pluc, Lodz
  - ETG Łódz, Lodz
  - Clinical Best Solutions Sp. Z O.O. Spółka Komandytowa, Lublin
  - Centrum Alergologii Teresa Hofman Sp. z o.o., Poznan
  - Specjalistyczna Przychodnia Lekarska ALERGO-MED Sp. z.o.o., Poznan
  - EMED Centrum Uslug Medycznych Ewa Śmiałek, Rzeszów
  - ETG Skierniewice, Skierniewice
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z.o.o, Tarnów
  - Specjalistyczne Centrum Medyczne Centermed Sp. z o.o., Tarnów
  - IRMED Irena Wojciechowska, Warsaw
  - WK Medical Service Sp. z o.o., Warsaw
  - "ALL-MED" Specjalistyczna Opieka Medyczna, Medyczny Instytut Badawczy, Wroclaw
  - Michał Bogacki - DOBROSTAN, Wroclaw
  - Niepubliczny Zakład Opieki Zdrowotnej Przychodnia Lekarska Hipokrates Sp. z o.o., Zabrze

REFERENCES:
- [Derived] Layhadi JA, Starchenka S, De Kam PJ, Palmer E, Wu LYD, Keane ST, Fulton WT, Hikmawati P, Meng X, Filipaviciute P, Cutrina Pons A, Oluwayi K, Lis K, Armfield O, Skinner MA, Heath MD, Hewings SJ, Kramer MF, Shamji MH. Modulation of Cellular, Molecular, and Humoral Responses by PQ Grass 27,600 SU for the Treatment of Seasonal Allergic Rhinitis: A Randomised Double Blind Placebo Control Exploratory Field Study. Allergy. 2026 Jan;81(1):232-247. doi: 10.1111/all.16640. Epub 2025 Jul 8. PMID 40626378

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PQ Grass | Placebo
Started | 278 | 277
Completed | 266 | 262
Not Completed | 12 | 15
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Sponsor request | 1 | 0
Not completed — Study terminated by Sponsor for site 202 moving to a different location | 3 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | PQ Grass | Placebo | Total
Number analyzed (Participants) | 278 | 277 | 555
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.02) | 34.8 (10.34) | 33.8 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 126 | 249
  Male | 155 | 151 | 306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 274 | 275 | 549
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 5 | 9
  White | 268 | 265 | 533
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Austria | 12 | 13 | 25
  Hungary | 1 | 0 | 1
  United States | 33 | 34 | 67
  Czechia | 34 | 33 | 67
  Poland | 77 | 76 | 153
  Germany | 121 | 121 | 242
Alcohol consumption [Count of Participants; unit: Participants] — Alcohol consumption was recorded as: never, currently daily, currently weekly, currently monthly currently occasionally, previously daily, previously weekly, previously monthly or previously occasionally
  Participants
    Never | 56 | 59 | 115
    Currently Daily | 3 | 6 | 9
    Currently Weekly | 30 | 29 | 59
    Currently Monthly | 29 | 26 | 55
    Currently Occasionally | 144 | 146 | 290
    Previously Daily | 1 | 0 | 1
    Previously Weekly | 1 | 1 | 2
    Previously Monthly | 8 | 7 | 15
    Previously Occasionally | 6 | 3 | 9
Smoking habit [Count of Participants; unit: Participants] — Smoking habit was recorded as: never, currently daily, currently weekly, currently monthly currently occasionally, previously daily, previously weekly, previously monthly or previously occasionally
  Participants
    Never | 209 | 204 | 413
    Currently Daily | 25 | 24 | 49
    Currently Weekly | 3 | 2 | 5
    Currently Monthly | 0 | 1 | 1
    Currently Occasionally | 9 | 16 | 25
    Previously Daily | 16 | 20 | 36
    Previously Weekly | 1 | 2 | 3
    Previously Monthly | 1 | 1 | 2
    Previously Occasionally | 14 | 7 | 21
Height [Mean (Standard Deviation); unit: cm] | 174.1 (9.70) | 173.7 (9.72) | 173.9 (9.70)
Weight [Mean (Standard Deviation); unit: Kg] | 80.44 (19.435) | 79.69 (17.327) | 80.07 (18.459)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI calculated as weight (kg)/height (m^2)
  Kg/m^2 | 26.45 (5.874) | 26.32 (5.018) | 26.39 (5.459)

OUTCOME MEASURES:

1. Primary Outcome: Combined Symptom and Medication Score (CSMS) Averaged Over the Peak Grass Pollen Season (GPS)
Description: The daily CSMS is calculated as the sum of the daily Symptom Score (dSS) and the daily Medication Score (dMS).
  The dSS component of the CSMS is calculated as the sum of 6 individual symptom (2 conjunctival and 4 nasal) scores, each with a range of 0 to 3 points and divided by 6, and therefore has a total range between 0 and 3.
  The dMS is a score assigned according to the step of relief medication used in a day (from 0: no relief medication to 3: oral corticosteroids with step and step 2 medications).
  The daily CSMS has a range between 0 and 6. The average CSMS over the peak GPS will be calculated as sum of the daily CSMS within the peak GPS divided by the number of days of the peak GPS where the CSMS has been collected. Higher values in the scale represent worse outcomes.
Time Frame: dSS and dMS are recorded daily between Visit 8 (wk 16-29) and Visit 11 (wk 28-41). Then CSMS is adjusted to the Peak GPS, which depends on the GPS start and end dates for each region
Population: Full analysis set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 278 | 277
score on a scale | 1.08 [0.84 to 1.30] | 1.34 [1.12 to 1.57]
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; Test type: Superiority; p = 0.00048, Mixed Models Analysis; relative difference (%) = -20.25, 95% CI 2-sided [-31.0 to -9.49]

2. Secondary Outcome: Combined Symptom and Medication Score (CSMS) Averaged Over the Entire (or Truncated) Grass Pollen Season (GPS)
Description: 6 individual symptoms assessed in a 4 point severity scale (0-No symptoms to 3-Severe symptoms) and combined with relief medication use assessed using a 4 point severity scale (0=No relief medication, 1=anti-histamine use, 2=nasal corticosteroid use, and 3=oral corticosteroid use)
Time Frame: dSS and dMS are recorded daily between Visit 8 (wk 16-29) and Visit 11 (wk 28-41). Then CSMS is adjusted to the entire GPS, which depends on the GPS start and end dates for each region
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 278 | 277
units on a scale | 0.99 (0.786) | 1.23 (0.965)
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; Test type: Superiority; p = 0.00032, Mixed Models Analysis; Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; relative difference (%) = -20.2, 95% CI 2-sided [-30.13 to -10.27]

3. Secondary Outcome: Daily Medication Score (dMS) Component of the CSMS Averaged Over the Peak GPS and Entire (or Truncated) GPS
Description: The dMS is calculated from the daily use of relief medication. Scores are assigned following the scheme:
  Score 0: no relief medication used Score 1: Oral antihistamine/Ocular antihistamine Score 2: Intranasal corticosteroid with Step 1 medication(s) Score 3: Oral corticosteroids with Step 1 and Step 2 medications The maximum dMS corresponds to a score of 3, which would indicate worse symptoms in the patient.
Time Frame: dMS of the CSMS was recorded daily between Visit 8 (wk 16-29) and Visit 11 (wk 28-41). Then dMS is adjusted to the peak or entire GPS
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 278 | 277
score on a scale
  dMS averaged over the peak GPS | 0.47 (0.554) | 0.59 (0.589)
  dMS averaged over the Entire (Truncated) GPS | 0.33 (0.393) | 0.46 (0.485)
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Comparison of dMS of CSMS on peak GPS; Test type: Superiority — Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; p = 0.00080, Mixed Models Analysis; relative difference (%) = -26.54, 95% CI 2-sided [-41.15 to -11.94]
Statistical Analysis 2: Comparison: PQ Grass vs Placebo; Comparison of dMS of CSMS on entire GPS; Test type: Superiority — Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; p = 0.00031, Mixed Models Analysis; relative difference (%) = -26.6, 95% CI 2-sided [-40.49 to -12.72]

4. Secondary Outcome: Daily Symptom Score (dSS) Component of the CSMS Averaged Over the Peak GPS and Entire (or Truncated) GPS
Description: dSS score is based on the sum of the score of 6 symptoms using a 4-point severity scale as follows: 0 = No symptoms
  1. = Mild symptoms
  2. = Moderate symptoms
  3. = Severe symptoms
  The dSS is calculated as the sum of the scores for the 6 individual symptoms, divided by 6. Higher values in the scale indicate worse symptoms.
Time Frame: dSS of the CSMS was recorded daily between Visit 8 (wk 16-29) and Visit 11 (wk 28-41). Then dMS is adjusted to the peak or entire GPS
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 278 | 277
score on a scale
  dSS averaged over peak GPS | 0.82 (0.589) | 0.95 (0.640)
  dSS Averaged Over the Entire (Truncated) GPS | 0.65 (0.478) | 0.78 (0.564)
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Comparison of dSS of CSMS on peak GPS; Test type: Superiority — Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; p = 0.00223, Mixed Models Analysis; relative difference (%) = -16.35, 95% CI 2-sided [-26.27 to -6.44]
Statistical Analysis 2: Comparison: PQ Grass vs Placebo; Comparison of dSS of CSMS on entire GPS; Test type: Superiority — Linear mixed model using treatment group as fixed effect and pooled geographical region as random effect; p = 0.00076, Mixed Models Analysis; relative difference (%) = -16.58

5. Secondary Outcome: Average Rhinoconjunctivitis Quality of Life Questionnaire With Standardized Activities (RQLQ(S)) Measured Within the Peak GPS
Description: RQLQ(S) is a health-related quality of life instrument that measures the functional impairments that are most troublesome to adults.
  It is measured in a 7-point scale (0 = not impaired at all - 6 = severely impaired) with higher scores reflecting a lower quality of life.
Time Frame: RQLQ(s) is performed at Visit 2 (wk 2-8), Visit 9 (wk 18-31) and Visit 10 (wk 23-36).
Population: FAS - RQLQ data was not available for all participants in the FAS. Number of subjects with RQLQ data is detailed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 137 | 123
score on a scale | 1.399 (1.0718) | 1.903 (1.2447)
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Average Total RQLQ Score During Peak GPS; Test type: Superiority; p = 0.00032, Mixed Models Analysis; Linear mixed model using treatment group as fixed effect, Baseline total RQLQ score as covariate and pooled geographical region as random effect; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.76 to -0.23]

6. Secondary Outcome: Change in Serum Grass-specific IgG4 (Immunoglobulin G4) From Baseline to Visit 7.
Description: Serum grass-specific IgG4 was measured at baseline and at visit 7
Time Frame: Serum grass-specific IgG4 was measured at Visit 1 (baseline) and Visit 7 (wk 12-25)
Population: FAS - IgG4 values were not available for all participants. Number of subjects with available data is detailed.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 229 | 243
mg/L | 3.95 [3.44 to 4.46] | -0.05 [-0.54 to .045]
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Change from baseline to Visit 7 of serum grass-specific IgG4 [mg/L]; Test type: Superiority; p < 0.00001, Mixed Models Analysis; Mean Difference (Final Values) = 3.99, 95% CI 2-sided [3.28 to 4.7]

7. Secondary Outcome: Number of Well Days During the Peak GPS
Description: A "well day" was defined based on CSMS as a day with:
  * No use of relief medication on the particular day, i.e., CSMS-dMS = 0;
  * And a total dSS, i.e., CSMS-dSS ≤ 2 out of 18 of the raw scores.
Time Frame: dMS and dSS was recorded daily between Visit 8 (wk 16-29) and Visit 11 (wk 28-41). Then number of well days was calculated during peak GPS.
Population: FAS - Determination of well days was not possible for all participants. Number of subjects with data available is detailed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 265 | 266
days | 6.6 (8.16) | 5.5 (7.11)
Statistical Analysis 1: Comparison: PQ Grass vs Placebo; Probability of Well Days During Peak (truncated) GPS; Test type: Superiority; p = 0.10846, Regression, Logistic; The probability of a well day was calculated using a generalized estimating equation (GEE) or similar approaches as appropriate; Odds Ratio (OR) = 1.254, 95% CI 2-sided [0.951 to 1.652]

8. Secondary Outcome: Frequency, Severity and Relationship of AEs (Adverse Event) to Treatment
Description: Number of subjects with at least one event of the specified AE type
Time Frame: From visit 1 (baseline) to last follow-up call (week 46)
Population: SAF - One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo. Safety results are based on treatment received.
Measure: Number; unit: number of subjects
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
number of subjects
  Total AEs | 232 | 163
  Definitely related AEs | 144 | 53
  Probably related AEs | 34 | 23
  Possibly related AEs | 34 | 31
  Unlikely related AEs | 1 | 4
  Not related AEs | 19 | 43

9. Secondary Outcome: Frequency of AEs Leading to Premature Discontinuation From Treatment or Clinical Trial
Description: Number of subjects with at least one event of the specified AE type
Time Frame: From visit 1 (baseline) to last follow-up call (week 46)
Population: as for outcome 8
Measure: Number; unit: number of subjects
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
number of subjects
  AE leading to premature discontinuation from treatment | 4 | 5
  AE leading to premature discontinuation from clinical trial | 1 | 3

10. Secondary Outcome: Frequency of AESI (Adverse Events of Special Interest)
Description: Number of subjects with at least one event of the specified AE type
Time Frame: From visit 1 (baseline) to last follow-up call (week 46)
Population: as for outcome 8
Measure: Number; unit: number of subjects
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
number of subjects | 0 | 0

11. Secondary Outcome: Changes in Serum Chemistry Values (Sodium, Potassium and Chloride) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: SAF - One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo. Safety results are based on treatment received. Serum chemistry was not available for all subjects, the number of available subjects for each analyte is detailed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 258 | 258
mmol/L
  Serum sodium change: number analyzed (Participants) | 257 | 258
  Serum sodium change | -0.1 (1.94) | -0.2 (1.85)
  Serum potassium change | -0.05 (0.464) | -0.04 (0.484)
  Serum chloride change: number analyzed (Participants) | 257 | 257
  Serum chloride change | 0.6 (2.04) | 0.3 (2.10)

12. Secondary Outcome: Changes in Serum Chemistry Values (Glucose, Uric Acid, Urea, Phosphorus and Cholesterol) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 259 | 260
mmol/L
  Serum glucose change | 0.065 (0.8844) | 0.142 (0.9704)
  Serum uric acid change: number analyzed (Participants) | 257 | 257
  Serum uric acid change | 0.005 (0.0427) | 0.009 (0.0466)
  Serum urea change: number analyzed (Participants) | 257 | 257
  Serum urea change | 0.36 (1.1356) | 0.28 (1.214)
  Serum total phosphorus change: number analyzed (Participants) | 257 | 255
  Serum total phosphorus change | 0.011 (0.2110) | 0.027 (0.1926)
  Serum total cholesterol change: number analyzed (Participants) | 257 | 257
  Serum total cholesterol change | -0.208 (0.6095) | -0.236 (0.6939)

13. Secondary Outcome: Changes in Serum Chemistry Values ( Calcium, Creatinine and Total Bilirubin) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 257 | 257
mmol/L
  Serum calcium change | -0.039 (0.0868) | -0.035 (0.0942)
  Serum creatinine change: number analyzed (Participants) | 228 | 229
  Serum creatinine change | 0.0022 (0.009517) | 0.0024 (0.00934)
  Serum total bilirubin change: number analyzed (Participants) | 256 | 254
  Serum total bilirubin change | 0.00029 (0.003945) | 0.00046 (0.004436)

14. Secondary Outcome: Changes in Serum Chemistry Values (Total Protein and Albumin) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 258 | 258
g/L
  Serum total protein change: number analyzed (Participants) | 257 | 258
  Serum total protein change | -2.0 (3.57) | -2.2 (3.66)
  Serum albumin change | -1.2 (2.46) | -1.0 (2.46)

15. Secondary Outcome: Changes in Serum Chemistry Values (Alkaline Phosphatase, Lactate Dehydrogenase, Aspartate Aminotransferase, Alanine Aminotransferase and Gamma-glutamyl Transferase) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 257 | 257
U/L
  Alkaline phosphatase | -2.5 (10.47) | -2.0 (10.86)
  Lactate dehydrogenase | 2.7 (23.11) | 4.2 (26.93)
  Aspartate aminotransferase: number analyzed (Participants) | 256 | 254
  Aspartate aminotransferase | 0.3 (15.51) | 1.3 (8.78)
  Alanine aminotransferase: number analyzed (Participants) | 256 | 254
  Alanine aminotransferase | -1.8 (20.73) | -0.9 (17.42)
  Gamma-glutamyl transferase | -0.5 (18.75) | -1.1 (9.09)

16. Secondary Outcome: Changes in Serum Chemistry Values (C-reactive Protein) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: SAF - One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo. Safety results are based on treatment received. Serum chemistry was not available for all subjects.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 257 | 260
mg/L | -0.33 (3.453) | -0.1 (3.991)

17. Secondary Outcome: Changes in Haematology Values (Red Blood Cells) Between Baseline and Visit 11
Description: The outcome includes total red blood cells number at visit 11 and change from baseline expressed as cells x 10^12/L
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: SAF - One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo. Safety results are based on treatment received. Serum chemistry was not available for all subjects, the number of available data for each analyte is detailed.
Measure: Mean (Standard Error); unit: number of cells(x10^12)/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 254 | 252
number of cells(x10^12)/L
  Absolute count of red blood cells at visit 11 | 4.81 (0.460) | 4.84 (0.465)
  Change in number of red blood cells from baseline to visit 11 | -0.03 (0.2242) | -0.03 (0.237)

18. Secondary Outcome: Changes in Hematology Values (White Blood Cells and Platelets) Between Baseline and Visit 11
Description: Outcomes include the change from baseline in the number of white blood cells and platelets expressed as cells x 10^9/L
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: number of cells(x10^9)/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 254 | 252
number of cells(x10^9)/L
  Change from baseline to visit 11 in the number of white blood cells | -0.21 (1.762) | -0.11 (1.469)
  Change from baseline to visit 11 in the number of platelets | -4.4 (60.00) | -12.5 (45.22)

19. Secondary Outcome: Change in Hematology Values (Hemoglobin) Between Baseline and Visit 11
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 254 | 252
g/L | -1.5 (7.75) | -1.4 (7.34)

20. Secondary Outcome: Changes in Clinical Laboratory Values (Urinalysis: pH) Between Baseline and Visit 11
Description: Urinalysis was performed using a urine dip-stick - Results were assessed by the investigators as clinical significant or not.
  The pH is measured in a scale from 0 to 14 (being 0 the most acid and 14 the most basic values)
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41).
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 257 | 256
units on a scale | -0.061 (1.0138) | 0.001 (1.0082)

21. Secondary Outcome: Clinical Laboratory Values (Urinalysis: Protein, Glucose, Bilirubin, Blood and Leukocytes) at Baseline and Visit 11
Description: Urinalysis was determined using a urine dip-stick - Results were scored as zero, traces, +1, +2, +3, +4 (being zero no detection of the parameter, and 4 the maximum value) Note: Microscopic examination was conducted if protein, leukocytes and/or blood are detected. If needed, microscopic examination included white blood cells, red blood cells, casts, and bacteria.
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
Participants
  Protein at screening: 0 | 264 | 257
  Protein at screening: Traces | 8 | 10
  Protein at screening: +1 | 5 | 7
  Protein at screening: +2 | 0 | 0
  Protein at screening: +3 | 0 | 0
  Protein at screening: +4 | 0 | 0
  Protein at screening: Missing | 2 | 2
  Protein at visit 11: 0 | 249 | 250
  Protein at visit 11: Traces | 6 | 5
  Protein at visit 11: +1 | 3 | 2
  Protein at visit 11: +2 | 1 | 1
  Protein at visit 11: +3 | 0 | 0
  Protein at visit 11: +4 | 0 | 0
  Protein at visit 11: Missing | 20 | 18
  Glucose at screening: 0 | 277 | 274
  Glucose at screening: Traces | 0 | 0
  Glucose at screening: +1 | 0 | 0
  Glucose at screening: +2 | 0 | 0
  Glucose at screening: +3 | 0 | 0
  Glucose at screening: +4 | 0 | 0
  Glucose at screening: Missing | 2 | 2
  Glucose at visit 11: 0 | 259 | 258
  Glucose at visit 11: Traces | 0 | 0
  Glucose at visit 11: +1 | 0 | 0
  Glucose at visit 11: +2 | 0 | 0
  Glucose at visit 11: +3 | 0 | 0
  Glucose at visit 11: +4 | 0 | 0
  Glucose at visit 11: Missing | 20 | 18
  Bilirubin at screening: 0 | 276 | 270
  Bilirubin at screening: Traces | 0 | 1
  Bilirubin at screening: +1 | 1 | 3
  Bilirubin at screening: +2 | 0 | 0
  Bilirubin at screening: +3 | 0 | 0
  Bilirubin at screening: +4 | 0 | 0
  Bilirubin at screening: Missing | 2 | 2
  Bilirubin at visit 11: 0 | 259 | 257
  Bilirubin at visit 11: Traces | 0 | 0
  Bilirubin at visit 11: +1 | 0 | 0
  Bilirubin at visit 11: +2 | 0 | 0
  Bilirubin at visit 11: +3 | 0 | 1
  Bilirubin at visit 11: +4 | 0 | 0
  Bilirubin at visit 11: Missing | 20 | 18
  Blood at screening: 0 | 261 | 264
  Blood at screening: Traces | 0 | 1
  Blood at screening: +1 | 5 | 3
  Blood at screening: +2 | 4 | 1
  Blood at screening: +3 | 4 | 1
  Blood at screening: +4 | 3 | 3
  Blood at screening: Missing | 2 | 3
  Blood at visit 11: 0 | 247 | 250
  Blood at visit 11: Traces | 3 | 1
  Blood at visit 11: +1 | 2 | 1
  Blood at visit 11: +2 | 4 | 0
  Blood at visit 11: +3 | 1 | 2
  Blood at visit 11: +4 | 2 | 4
  Blood at visit 11: Missing | 20 | 18
  Leukocytes at screening: 0 | 263 | 252
  Leukocytes at screening: Traces | 3 | 0
  Leukocytes at screening: +1 | 3 | 2
  Leukocytes at screening: +2 | 3 | 3
  Leukocytes at screening: +3 | 4 | 1
  Leukocytes at screening: +4 | 1 | 0
  Leukocytes at screening: Missing | 2 | 18

22. Secondary Outcome: Clinical Laboratory Values (Urinalysis: Ketones, Nitrite, Urobilinogen ) at Baseline and Visit 11
Description: Urinalysis was performed using a urine dip-stick - Results were represented as negative or positive Note: Microscopic examination was conducted if nitrite was detected. If needed, microscopic examination included white blood cells, red blood cells, casts, and bacteria.
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo. Safety results are based on treatment received.
  Serum chemistry was not available for all subjects, the number of available data for each analyte is detailed.
Measure: Count of Participants; unit: Participants
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
Participants
  Ketones at screening: Negative | 277 | 273
  Ketones at screening: Positive | 0 | 1
  Ketones at screening: Missing | 2 | 2
  Ketones at visit 11: Negative | 257 | 257
  Ketones at visit 11: Positive | 2 | 1
  Ketones at visit 11: Missing | 20 | 18
  Nitrite at baseline: Negative | 274 | 272
  Nitrite at baseline: Positive | 3 | 2
  Nitrite at baseline: Missing | 2 | 2
  Nitrite at visit 11: Negative | 257 | 258
  Nitrite at visit 11: Positive | 2 | 0
  Nitrite at visit 11: Missing | 20 | 18
  Urobilinogen at screening: Negative | 277 | 274
  Urobilinogen at screening: Positive | 0 | 0
  Urobilinogen at screening: Missing | 2 | 2
  Urobilinogen at visit 11: Negative | 259 | 257
  Urobilinogen at visit 11: Positive | 0 | 1
  Urobilinogen at visit 11: Missing | 20 | 18

23. Secondary Outcome: Changes in Vital Signs (Systolic and Diastolic Blood Pressure) From Baseline to All Treatment Visits
Description: Blood pressure was measured (in millimeters of mercury) at all treatment visits: Visit (V)1, V2 (2-8 weeks), V3 (3-9 weeks), V4 (4-10 weeks), V5 (7-15 weeks), V6 (10-20 weeks), V7 (week 13-25), V8 (16.29 weeks), V9 (18-31 weeks), V10 (23-36 weeks), V11 (28-41 weeks). At Visits 2 to 7, vital sign measurements were performed before and 30 to 60 minutes following investigational drug/placebo administration.
Time Frame: From Visit 1 (baseline) to visit 11 (week 28-41)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PQ Grass | Placebo
Number analyzed (Participants) | 279 | 276
mmHg
  Systolic blood pressure at visit 2 (post-dose) - Baseline | -1.2 (7.93) | -1.5 (7.97)
  Systolic blood pressure at visit 3 (pre-dose) - Baseline: number analyzed (Participants) | 276 | 273
  Systolic blood pressure at visit 3 (pre-dose) - Baseline | 0.4 (9.22) | 0.00 (9.32)
  Systolic blood pressure at visit 3 (post-dose) - Baseline: number analyzed (Participants) | 276 | 273
  Systolic blood pressure at visit 3 (post-dose) - Baseline | -1.8 (9.75) | -1.4 (9.74)
  Systolic blood pressure at visit 4 (pre-dose) - Baseline: number analyzed (Participants) | 269 | 268
  Systolic blood pressure at visit 4 (pre-dose) - Baseline | 0.3 (10.29) | 0.4 (10.33)
  Systolic blood pressure at visit 4 (post-dose) - Baseline: number analyzed (Participants) | 269 | 268
  Systolic blood pressure at visit 4 (post-dose) - Baseline | -1.1 (9.94) | -2.1 (10.05)
  Systolic blood pressure at visit 5 (pre-dose) - Baseline: number analyzed (Participants) | 266 | 265
  Systolic blood pressure at visit 5 (pre-dose) - Baseline | 0.6 (10.06) | -0.7 (10.07)
  Systolic blood pressure at visit 5 (post-dose) - Baseline: number analyzed (Participants) | 266 | 265
  Systolic blood pressure at visit 5 (post-dose) - Baseline | -1.7 (9.28) | -2.3 (10.45)
  Systolic blood pressure at visit 6 (pre-dose) - Baseline: number analyzed (Participants) | 264 | 262
  Systolic blood pressure at visit 6 (pre-dose) - Baseline | -0.3 (10.06) | -0.3 (10.29)
  Systolic blood pressure at visit 6 (post-dose) - Baseline: number analyzed (Participants) | 263 | 262
  Systolic blood pressure at visit 6 (post-dose) - Baseline | -2.0 (10.52) | -2.3 (10.69)
  Systolic blood pressure at visit 7 (pre-dose) - Baseline: number analyzed (Participants) | 252 | 256
  Systolic blood pressure at visit 7 (pre-dose) - Baseline | -0.7 (10.10) | -1.9 (10.65)
  Systolic blood pressure at visit 7 (post-dose) - Baseline: number analyzed (Participants) | 251 | 255
  Systolic blood pressure at visit 7 (post-dose) - Baseline | -2.5 (10.12) | -3.0 (10.51)
  Systolic blood pressure at visit 8 - Baseline: number analyzed (Participants) | 269 | 266
  Systolic blood pressure at visit 8 - Baseline | -1.4 (10.04) | -1.1 (10.40)
  Systolic blood pressure at visit 9 - Baseline: number analyzed (Participants) | 269 | 264
  Systolic blood pressure at visit 9 - Baseline | -0.5 (10.66) | -1.9 (10.45)
  Systolic blood pressure at visit 10 - Baseline: number analyzed (Participants) | 267 | 262
  Systolic blood pressure at visit 10 - Baseline | -0.9 (11.12) | -1.8 (10.78)
  Systolic blood pressure at visit 11 - Baseline | -1.2 (11.07) | -2.3 (11.11)
  Diastolic blood pressure at visit 2 (post-dose) - Baseline | 0.2 (5.77) | -0.1 (6.70)
  Diastolic blood pressure at visit 3 (pre-dose) - Baseline: number analyzed (Participants) | 276 | 273
  Diastolic blood pressure at visit 3 (pre-dose) - Baseline | -0.2 (7.48) | -0.4 (7.52)
  Diastolic blood pressure at visit 3 (post-dose) - Baseline: number analyzed (Participants) | 276 | 273
  Diastolic blood pressure at visit 3 (post-dose) - Baseline | -1.0 (7.00) | -0.7 (8.00)
  Diastolic blood pressure at visit 4 (pre-dose) - Baseline: number analyzed (Participants) | 269 | 268
  Diastolic blood pressure at visit 4 (pre-dose) - Baseline | 0.2 (7.43) | -0.4 (7.67)
  Diastolic blood pressure at visit 4 (post-dose) - Baseline: number analyzed (Participants) | 269 | 265
  Diastolic blood pressure at visit 4 (post-dose) - Baseline | -0.7 (7.91) | -1.1 (7.73)
  Diastolic blood pressure at visit 5 (pre-dose) - Baseline: number analyzed (Participants) | 266 | 265
  Diastolic blood pressure at visit 5 (pre-dose) - Baseline | -0.1 (7.93) | -0.6 (8.05)
  Diastolic blood pressure at visit 5 (post-dose) - Baseline: number analyzed (Participants) | 266 | 265
  Diastolic blood pressure at visit 5 (post-dose) - Baseline | -0.3 (7.93) | -1.3 (8.37)
  Diastolic blood pressure at visit 6 (pre-dose) - Baseline: number analyzed (Participants) | 264 | 262
  Diastolic blood pressure at visit 6 (pre-dose) - Baseline | -0.5 (7.68) | 0.2 (7.91)
  Diastolic blood pressure at visit 6 (post-dose) - Baseline: number analyzed (Participants) | 263 | 262
  Diastolic blood pressure at visit 6 (post-dose) - Baseline | -0.7 (7.76) | -1.4 (7.91)
  Diastolic blood pressure at visit 7 (pre-dose) - Baseline: number analyzed (Participants) | 252 | 256
  Diastolic blood pressure at visit 7 (pre-dose) - Baseline | -0.5 (8.09) | -0.7 (8.54)
  Diastolic blood pressure at visit 7 (post-dose) - Baseline: number analyzed (Participants) | 251 | 255
  Diastolic blood pressure at visit 7 (post-dose) - Baseline | -0.7 (7.77) | -1.3 (8.52)
  Diastolic blood pressure at visit 8 - Baseline: number analyzed (Participants) | 269 | 266
  Diastolic blood pressure at visit 8 - Baseline | -1.4 (8.08) | -0.9 (8.25)
  Diastolic blood pressure at visit 9 - Baseline: number analyzed (Participants) | 269 | 264
  Diastolic blood pressure at visit 9 - Baseline | -0.4 (8.19) | -1.8 (7.72)
  Diastolic blood pressure at visit 10 - Baseline: number analyzed (Participants) | 267 | 262
  Diastolic blood pressure at visit 10 - Baseline | -0.3 (8.12) | -0.9 (8.56)
  Diastolic blood pressure at visit 11 - Baseline: number analyzed (Participants) | 266 | 263
  Diastolic blood pressure at visit 11 - Baseline | -0.1 (8.42) | -1.3 (8.88)

ADVERSE EVENTS:
Time Frame: AE were reported throughout the study from visit 1 (baseline) to the last follow-up call (week 40-46)
Description: One subject randomized to placebo received PQ Grass throughout the trial, consequently 279 subjects were treated with PQ Grass and 276 subjects with placebo; results are based on treatment received
Arm/Group | PQ Grass | Placebo
All-Cause Mortality (participants affected / at risk) | 0/279 | 0/276
Serious Adverse Events (participants affected / at risk) | 5/279 | 3/276
Other Adverse Events (participants affected / at risk) | 226/279 | 155/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PQ Grass (N=279) | Placebo (N=276)
anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Rhythm idioventricular (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PQ Grass (N=279) | Placebo (N=276)
Headache (Nervous system disorders) | 26 | 20
Injection site erythema (General disorders) | 183 | 28
Injection site swelling (General disorders) | 161 | 43
Injection site pain (General disorders) | 123 | 65
Injection site pruritus (General disorders) | 133 | 24
Injection site warmth (General disorders) | 19 | 5
Injection site urticaria (General disorders) | 16 | 1
Eye pruritus (Eye disorders) | 23 | 23
Lacrimation increased (Eye disorders) | 14 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 35 | 25
Sneezing (Respiratory, thoracic and mediastinal disorders) | 34 | 27
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 | 26
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 16 | 23
Nasopharyngitis (Infections and infestations) | 28 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT05540717/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT05540717/SAP_003.pdf